CLINICAL TRIAL: NCT02672319
Title: Endoscopic Ultrasound (EUS) Guided Cyanoacrylate Injection for Variceal Obturation as Secondary Prophylaxis for Patients at High Risk for Recurrent Gastroesophageal Variceal Bleeding
Brief Title: EUS-guided Glue Injection for Varices Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond Shing Yan Tang, Clinical Professional Consultant, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EUS Glue Study
Record Dates: First submitted 2015-09-09; First posted 2016-02-03 (Estimated); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Gastroesophageal Varices

STUDY DESIGN:
Intervention Model Description: Comparison of clinical outcomes of a prospective study cohort to those in a historical control group
Oversight: Data Monitoring Committee: No

ARMS (2):
- EUS-guided glue injection (Experimental): Gastroesophageal varices > 3mm in diameter will be treated with EUS guided cyanoacrylate injection for variceal obturation in standard fashion. A conventional 19G needle (19G-Echotip needle, Cook Medical, USA) will be advanced into the target varix under real-time EUS guidance. Cyanoacrylate injection (Histoacryl, B. Braun Surgical, Germany) will be performed according to established protocol. Each aliquot of cyanoacrylate injection will consist of 0.5ml of Histoacryl + 0.7ml of lipiodol. 1 - 3 aliquots of cyanoacrylate injection may be given depending on the number of varices needed to be treated. EUS with colour Doppler will be used to monitor obliteration of blood flow in varices during and after cyanoacrylate injection.
  Interventions: Procedure: EUS-guided glue injection
- Historical control (No Intervention): A historical control group of HCC patients with gastroesophageal variceal bleeding who underwent conventional cyanoacrylate injection by OGD for index variceal bleeding based on de-identified data from an existing prospective GI bleed database from 2009-2013 would also be included to allow a more meaningful interpretation of the rebleeding rate from gastroesophageal varices from this study.

INTERVENTIONS:
Procedure: EUS-guided glue injection — Experimental: EUS-guided glue injection Gastroesophageal varices > 3mm in diameter will be treated with EUS guided cyanoacrylate injection for variceal obturation in standard fashion. A conventional 19G needle (19G-Echotip needle, Cook Medical, USA) will be advanced into the target varix under real-time EUS guidance. Cyanoacrylate injection (Histoacryl, B. Braun Surgical, Germany) will be performed according to established protocol. Each aliquot of cyanoacrylate injection will consist of 0.5ml of Histoacryl + 0.7ml of lipiodol. 1 - 3 aliquots of cyanoacrylate injection may be given depending on the number of varices needed to be treated. EUS with colour Doppler will be used to monitor obliteration of blood flow in varices during and after cyanoacrylate injection.
  Arms: EUS-guided glue injection

SUMMARY:
Bleeding from gastroesophageal varices is one of the major complications of cirrhosis. After successful treatment of the acute bleeding episode, patients who do not receive follow-up treatment to prevent rebleeding were reported to have a rebleeding rate of 60% within 1- 2 years. The presence of liver cancer and/or portal vein thrombosis has been associated with recurrent variceal bleeding. In a study of liver cancer patients in Hong Kong, 7.9% of patients developed at least 1 episode of variceal bleeding over the course of liver cancer.

In patients with portal hypertension from cirrhosis, current guidelines recommend non-selective beta-blocker, endoscopic band ligation for esophageal varices after initial bleeding, and either cyanoacrylate injection for variceal obturation or transjugular intrahepatic portosystemic shunt for gastric varices after initial bleeding. However, it is unclear whether the above strategies will have the same clinical effect for patients with liver cancer and/or portal vein thrombosis who are at high risk for recurrent bleeding.

Recently, the technique of endoscopic ultrasound (EUS) guided cyanoacrylate (glue) injection for variceal obturation has been described. In a study of patients with gastric variceal bleeding, EUS guided glue injection and coiling was reported to achieve hemostasis in all patients and 96% of the gastric varices remained obliterated during the follow-up period. To date, there has been no dedicated study to evaluate the role of EUS guided glue injection for prevention of future bleeding in patients at high risk for recurrent variceal bleeding such as those with liver cancer or portal vein thrombosis.

The investigators propose this study to evaluate the feasibility and safety of EUS guided glue injection for follow-up variceal treatment in patients at high risk for recurrent variceal bleeding, such as those with liver cancer and/or portal vein thrombosis.

DETAILED DESCRIPTION:
Gastroesophageal variceal bleeding is one of the major complications of cirrhosis and occurs at a rate of 5 to 15% per year. 50% of patients with cirrhosis develop variceal bleeding during their lifetime. Large varix size, presence of red wale signs on endoscopy, and decompensated cirrhosis are predictors of variceal hemorrhage. Current first-line management of acute variceal bleeding includes a combination of vasoactive drug, endoscopic therapy and antibiotic prophylaxis. Despite advances in the management of acute variceal bleeding, the 6-week mortality remains significant at 15 - 20% per episode of variceal bleeding.

In patients who survive the acute variceal bleeding episode but without secondary prophylaxis, the median rebleeding rate is about 60% within 1- 2 years of the index bleeding with a mortality of 33%. The presence of hepatocellular carcinoma (HCC) and/or portal vein thrombosis (PVT) have been associated with recurrent variceal bleeding and worse outcome. In a retrospective study of 2928 HCC patients in Hong Kong, 7.9% of the patients developed at least 1 episode of variceal bleeding over the course of HCC. In cirrhotic patients with PVT but without HCC, variceal bleeding is not an uncommon complication.

In patients with portal hypertension from cirrhosis, current guidelines recommend non-selective beta-blocker, endoscopic band ligation for esophageal varices after initial bleeding, and either cyanoacrylate injection for variceal obturation or transjugular intrahepatic portosystemic shunt for gastric varices after initial bleeding. However, it is unclear whether the above strategies will have the same clinical effect for patients with liver cancer and/or portal vein thrombosis who are at high risk for recurrent bleeding.

Recently, the technique of endoscopic ultrasound (EUS) guided cyanoacrylate (glue) injection for variceal obturation has been described. In a study of patients with gastric variceal bleeding, EUS guided glue injection and coiling was reported to achieve hemostasis in all patients and 96% of the gastric varices remained obliterated during the follow-up period. To date, there has been no dedicated study to evaluate the role of EUS guided glue injection for prevention of future bleeding in patients at high risk for recurrent variceal bleeding such as those with liver cancer or portal vein thrombosis.

The investigators propose this study to evaluate the feasibility and safety of EUS guided glue injection for follow-up variceal treatment in patients at high risk for recurrent variceal bleeding, such as those with liver cancer and/or portal vein thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with hepatocellular carcinoma (liver cancer), and/or portal vein thrombosis, who have presented with gastroesophageal variceal bleeding within 12 weeks
* Age > 18 years
* Written informed consent available

Exclusion Criteria:

* Contraindications for endoscopy due to comorbidities
* Unable to provide written informed consent
* Refractory coagulopathy (INR>1.5) or refractory thrombocytopenia (platelets <50,000) despite blood product transfusion
* Pregnant patients
* Moribund patients from terminal illnesses

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Rebleeding rate | 6 months
  Number of participants who undergo EUS guided glue injection and develop rebleeding during the 3-month and 6-month follow up period

SECONDARY OUTCOMES:
bleeding free interval after index procedure | 12 months
  Duration without bleeding from varices
Technical success | At time of procedure
  Technical success = successful delivery of glue injection under EUS guidance
procedural complication | 12 months
  Procedure related complication such as perforation, bleeding, infection, cardiopulmonary adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Raymond S Tang, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No